CLINICAL TRIAL: NCT03264365
Title: The Effectiveness of a Post-ICU Recovery Program on Relatives to Patients Receiving Mechanically Ventilatory Support: Data Linked to RAPIT-I Investigation
Brief Title: The Effectiveness of a Post-ICU Recovery Program on Relatives
Acronym: RAPIT-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Collaborators: Nordsjaellands Hospital (Other); Herlev Hospital (Other); Horsens Hospital (Other); Nykøbing Falster County Hospital (Other); Naestved Hospital (Other); Rigshospitalet, Denmark (Other); Aabenraa Hospital (Other); Sonderborg Hospital (Other Government); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Svendborg Hospital (Other)
Responsible Party: Principal Investigator, Janet Froulund Jensen, PHD, Holbaek Sygehus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01863 HIH-2012-011; NCT-01721239 (Other: Registry Identifier of RAPIT-I on ClinicalTrials.gov)
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Intensive Care Unit Syndrome; Relatives
Keywords: Health-related quality of life; Anxiety; Depression; Post-traumatic stress disorder; Recovery programme; Rehabilitation; Follow-up programme; Aftercare; Randomized controlled Trial; Multicentre
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic | interventions — Methods; Standard of Care

STUDY DESIGN:
Intervention Model Description: Pragmatic, non-blinded, multicenter, parallel-group randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Data analyses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Relatives participated actively in the one out of three consultation conducted by trained study nurses at two months after intensive care superimposed on standard care.
  Interventions: Behavioral: Intervention
- Standard care (No Intervention): Relatives to former ICU patients, who had received standard care (SC) completed a questionnaire package at 3 and 12 months after the patient was discharged from intensive care. After enrollment were all contract handled by primary investigator.

INTERVENTIONS:
Behavioral: Intervention — Intervention (plus standard care)
  * Patients photographs during the ICU-stay,
  * Written information about life after ICU
  * First consultation face-to-face in hospital setting at three months after ICU
  * Visit ICU and photographs given
  * Consultations as needed
  Other Names: Standard care
  Arms: Intervention

SUMMARY:
Relatives of intensive care patients are at risk of developing symptoms of anxiety, depression and post-traumatic stress disorder resulting in impaired health-related quality of life (HRQOL). Recovery programs have been tested, but its effectiveness is sparse. The hypothesis is that relatives to former intensive care patients will improve their HRQOL one year after intensive care. We want to determine whether relatives to former intensive care patient's benefits from a recovery programme with improved HRQOL, Sense Of Coherence (SOC) and symptoms of anxiety, depression and PTSD compared to standard care one year after intensive care.

DETAILED DESCRIPTION:
Relatives of intensive care patients are affected of critical illness with symptoms of anxiety, depression and post-traumatic stress disorder resulting in impaired mental health. Recovery programs aimed at patients after a stay at the intensive care unit (ICU) have been tested and implemented, but the effectiveness is inconclusive, and on relatives sparse. The aim is to determine whether relatives to former intensive care patients benefits from a recovery programme with improved health-related quality of life (HRQOL), Sense Of Coherence (SOC), and symptoms of anxiety, depression, and PTSD compared to standard care during the first year after ICU discharge.

This was a sub-study of the "Recovery and Aftercare in Post-Intensive care Therapy patients" (RAPIT) trial; a pragmatic, non-blinded, multicentre, parallel-group, randomized controlled trial. We recruited patients and relatives concurrently during the RAPIT-trial study-period, and now we are doing analysis on relatives. We wants to include adult relatives defined by the patients from 10 Danish ICUs.

The study was powered to detect an effect size of a 5-point increase in the Medical Health Survey Short-Form 36 (SF-36) on the mental component score (MCS) in the intervention group at 12 months post-ICU. Power calculation was based on an expected distribution of MCS from a matched population with a mean of 36.7 (SD 11.7) from a similar study. With a statistical power of 80% and significance level of 0.05, we estimated that 86 relatives were needed in each group to complete follow-up.

The statistical analysis plan was based on intention-to-treat (ITT) as was per protocol (PP) analysis and investigating difference between intervention and controls. Relatives were considered to have received the intervention if the patient attended at least one of the three consultations, which accounted for the PP analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Defined by the patients

Exclusion Criteria:

* If the patients dropped out or died during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2012-12-15 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Mental Component Score | 12 months after ICU
  Health-related Quality of life using Short-form-36 questionnaire

SECONDARY OUTCOMES:
Mental Component Score | 3 months after ICU
  Health-related Quality of life using Short-form-36 questionnaire
Physical Component Score | 3 months after ICU
  Health-related Quality of life using Short-form-36 questionnaire
Physical Component Score | 12 months after ICU
  Health-related Quality of life using Short-form-36 questionnaire
Anxiety | 3 months after ICU
  Anxiety measured by Hospital Anxiety and Depression Scale (HADS)
Anxiety | 12 months after ICU
  Anxiety measured by Hospital Anxiety and Depression Scale (HADS)
Depression | 3 months after ICU
  Depression measured by Hospital Anxiety and Depression Scale (HADS)
Depression | 12 months after ICU
  Depression measured by Hospital Anxiety and Depression Scale (HADS)
Post-traumatic stress Disorders | 3 months after ICU
  Post-traumatic stress measured by the Harvard trauma Quesionnaire, ver. IV
Post-traumatic stress Disorders | 12 months after ICU
  Post-traumatic stress measured by the Harvard trauma Quesionnaire, ver. IV
Sense of coherence | 3 months after ICU
  Sense Of Coherence measured by the 13-item Orientation to Life questionnaire Questionnaire
Sense of coherence | 12 months after ICU
  Sense Of Coherence measured by the 13-item Orientation to Life questionnaire Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: RAPIT Steering Committee, Study Chair — Region of Copenhagen Capital and Region of Zealand
Locations (1):
- Holbæk Hospital, Holbæk, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Agreement of collaboration between sites have determinated that abstracts should be evaluated by the RAPIT-steering committee prior data are shared with other researchers.

REFERENCES:
- [Background] Jensen JF, Egerod I, Bestle MH, Christensen DF, Elklit A, Hansen RL, Knudsen H, Grode LB, Overgaard D. A recovery program to improve quality of life, sense of coherence and psychological health in ICU survivors: a multicenter randomized controlled trial, the RAPIT study. Intensive Care Med. 2016 Nov;42(11):1733-1743. doi: 10.1007/s00134-016-4522-1. Epub 2016 Sep 30. PMID 27695894